CLINICAL TRIAL: NCT03172039
Title: Antimicrobial Use and Stewardship in an Outpatient Hemodialysis Unit
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Marisa Battistella, Clinician Scientist, University Health Network, Toronto
Other Study IDs: 16-6388
Record Dates: First submitted 2017-05-28; First posted 2017-06-01 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: End Stage Renal Failure on Dialysis; Infection, Bacterial
Keywords: hemodialysis; antimicrobial stewardship; antimicrobial agents; bacterial infections; ambulatory care
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This quality improvement study will assess the antimicrobial use and prescribing practices of hospital and community prescribers for the ambulatory hemodialysis (HD) population in an urban academic outpatient HD unit in Ontario. Currently, in the outpatient HD unit at Toronto General Hospital (TGH), it is the standard of care for the patients to be screened on a weekly basis by the nephrology care team for the use of any oral or intravenous antimicrobials. Patient charts, pharmacy patient profiles and electronic medical records for these patients from September 1 2016 - April 30 2017 will be retrospectively reviewed in order to characterize antimicrobial use and its concordance with available clinical guidelines and antimicrobial stewardship principles described by the Centers for Disease Control and Prevention (CDC). The primary objective of the study is to determine the prevalence of antimicrobial use in an ambulatory HD population. The secondary objective of the study is to determine the congruence of prescribed antimicrobial regimens with available clinical guidelines and antimicrobial stewardship principles described by the CDC. It is hypothesized that antimicrobial use among HD patients will be common and that antimicrobial prescribing practices are not congruent with recommendations from published clinical guidelines and antimicrobial stewardship principles for a significant proportion of patients included in the retrospective review. Descriptive analysis of the data will summarize the findings. Future research will build upon the results of this project, and may include the development of interventions that target gaps in knowledge and prescribing behaviours of prescribers who provide care to the ambulatory HD population.

DETAILED DESCRIPTION:
Description of Study:

Patients who make up the ambulatory hemodialysis (HD) population at Toronto General Hospital (TGH) are interviewed on a weekly basis about their antimicrobial use during the nursing-led bedside huddle as part of the standard of care. These huddles take place daily during each of the four HD shifts: morning, afternoon, evening and nocturnal. During the huddle the nurse or patient care coordinator asks the patient if they have been prescribed an oral or intravenous antimicrobial by a hospital or community prescriber in the past 7 days. A Best Possible Medication History (BPMH) is completed by a HD Pharmacy team member for all patients who stated they have started a new antimicrobial. A BPMH is a patient's medication history which is defined as "a systematic process of interviewing the patient/family", and "a review of at least one other reliable source of information" (e.g., dispensing pharmacy records, hospital discharge records etc.) to confirm medication use. The BPMH is part of routine care in the HD unit and obtained at regular intervals (e.g., when a medication is started, changed or discontinued) to ensure the most accurate medication history is available. The BPMH containing information about the antimicrobial treatment is documented in the patient's medical chart, as well as in the electronic pharmacy patient profile. There will be no disruption to the current pharmacy practice and workflow in the HD unit by this study.

At the end of the data collection period, a panel compromising of a pharmacy resident, antimicrobial stewardship pharmacist, nephrology pharmacist, nurse practitioner and nephrologist will adjudicate each antimicrobial prescription with a presumed indication for congruence with available clinical guidelines and antimicrobial principles described by CDC. Each antimicrobial regimen will be categorized as congruent or non-congruent; any regimen for which there is inadequate or unavailable documentation in support of congruence will be classified as unknown congruence. The primary tool for assessing antimicrobial therapy will be against antimicrobial stewardship best practices guiding principles established by CDC, supplemented by applicable guidelines for each site of suspected infection published by major infectious disease and nephrology societies. Evidence-based resources for drug dosing in renal failure will be used to determine whether the prescribed antimicrobial regimen is consistent with literature-based dosing recommendations. The prescription will be assessed for types of stewardship-discordant prescribing that will be defined based on general stewardship principles a priori such as the following:

i) antimicrobial regimen has incorrect dose/route/frequency for intended infectious syndrome, pathogens and/or patient factors ii) length of treatment too short (discontinuation before adequate source control or clinical stability) or too long (prolonged therapy despite documented microbiologic clearance or resolution of symptoms) iii) empiric therapy spectrum too broad or narrow considering possible causative pathogens iv) antimicrobial therapy not tailored/streamlined/de-escalated for microbiology results v) non-infectious syndrome

Number of subjects:

The outpatient HD unit at TGH has a typical census of 300 patients. It is estimated that approximately 300 patient charts will be identified for inclusion as this study will be a non-comparative analysis of all patients admitted to the HD unit.

Statistics:

Data will be tabulated and analyzed using Microsoft Excel software. Descriptive statistics will be used to analyze the data. Means and standard deviations, as well as counts and proportions will be calculated for baseline parameters and relevant endpoints as appropriate. No interim analyses of the data are anticipated.

Procedure for accounting for missing, unused, and spurious data:

A patient's medical chart and pharmacy patient profile are comprehensive for obtaining a patient's medication history and therefore missing data should not be a concern. If this issue arises all available data sources will be exhausted (e.g., electronic patient record, pharmacy patient profiles).

Quality Assurance:

All data will be collected by the designated study team member using a data collection sheet and following a systematic approach approved by the project team. Raw data will be validated and reviewed by the project team following the completion of data collection and prior to data analysis.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Receiving outpatient hemodialysis (HD) for at least 3 months
* Prescribed at least one oral or intravenous antimicrobial (antibacterial or antifungal or antiviral) by a hospital or community prescriber between September 2016 to April 30 2017 inclusive

Exclusion Criteria:

* In-patients admitted to hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population to be studied in this retrospective chart review includes patients with end-stage renal disease receiving outpatient hemodialysis (HD) treatment at Toronto General Hospital (TGH) who were prescribed at least one antimicrobial during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of antimicrobial prescriptions in an ambulatory hemodialysis population | September 1 2016 - April 30 2017
  Prevalence will be determined by the total number of antimicrobial prescriptions in the study population over the period of study. An antimicrobial prescription will be defined as any oral or intravenous antibacterial or antifungal or antiviral agent prescribed by a community or hospital prescriber to a patient receiving hemodialysis (HD) from Toronto General Hospital's outpatient HD unit. An antimicrobial prescription will follow the 21-day rule.The 21-day rule is that there must be 21 or more days from the end of one antimicrobial course to the beginning of a second antimicrobial course for two courses to be reported as separate prescriptions. If antimicrobials are stopped for fewer than 21 days and then restarted, the second start is not considered a new prescription, and therefore will not be reported.

SECONDARY OUTCOMES:
Congruence of prescribed antimicrobial regimens | September 1 2016 - April 30 2017
  Proportion of antimicrobial prescriptions congruent with available clinical guidelines and antimicrobial stewardship principles based on:
  i) indication ii) antimicrobial agent iii) spectrum of activity against most likely causative pathogen iv) dose v) route of administration vi) dosing frequency vii) length of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No